CLINICAL TRIAL: NCT06108973
Title: Evaluation of Consumption of Sevoflurane in Chronic Obstructive Pulmonary Disease Patients Under General Anesthesia
Brief Title: Evaluation of Consumption of Sevoflurane in Chronic Obstructive Pulmonary Disease Patients
Acronym: SevoCOPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Employee's State Insurance Corporation, New Delhi (Other Government)
Collaborators: Medtronic Spine LLC (Industry)
Responsible Party: Principal Investigator, Santhosh Kumar T N, Nursing Orderly, Employee's State Insurance Corporation, New Delhi
Other Study IDs: 00127102023
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Capnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Normal Patients: Normal patients without any Lung Pathology for General Anesthesia
  Interventions: Device: Capnography
- COPD patients: Established Chronic Obstructive Pulmonary Disease for General Anesthesia
  Interventions: Device: Capnography

INTERVENTIONS:
Device: Capnography — To know the Co2 graph in COPD and Normal patients under General Anesthesia

SUMMARY:
All the Patients undergoing General Anesthesia and the patients who are having Chronic Obstructive Pulmonary Disease will be considered for this study. The Volume consumption of Sevoflurane will be studied in accordance with age, sex, duration , type of surgery, site of surgery and BMI.The volume consumption of sevoflurane is compared with Chronic Obstructive Pulmonary Disease and Normal Patients .

DETAILED DESCRIPTION:
Chronic Obstructive pulmonary disease is known to escalate the consumption of Inhalation Agents in General Anesthesia. Hence the Data to Collect the Official Record

ELIGIBILITY:
Inclusion Criteria:

* Both Sex All Age Group Patient willing to give consent COPD patient

Exclusion Criteria:

* Not willing to give consent Cancerous Lung Lung Lobectomy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Geography South East Asia-Sothern Peninsular INDIA'
  Soci Economic Mid Earning
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Estimation of Volume consumption of Sevoflurane | 8 weeks
  The consumption is expressed in Volume ml/kg

CONTACTS AND LOCATIONS:
Overall Officials: Dr Manjunath, MD, Principal Investigator — ESIC

IPD SHARING:
Plan to Share IPD: No